CLINICAL TRIAL: NCT03406143
Title: Evaluation of the Effect of CGF in Promoting Mechanical-stretch Induced in Vivo Skin
Brief Title: Evaluation of the Effect of CGF in Promoting Mechanical-stretch Induced in Vivo Skin Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, M.D., Ph.D.,Head of PRS Department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGFskin
Record Dates: First submitted 2017-12-19; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGF injection group (Experimental): Concentrate Growth Factors(CGF) will be harvested through centrifugation afte intravenous blood collection. Venous blood was collected in tube and then centrifuged in Medifuge system（Thermo Scientific）. About 2ml liquid CGF can be harvested from 9ml venous blood. Patients will receive autologous CGF injection subdermally to expanded skin at the density of 0.02 ml/cm2.
  Interventions: Procedure: CGF injection
- Control group (Sham Comparator): 0.9% saline will be injected into expanded skin for control study. Patients will receive saline injection subdermally to expanded skin at the density of 0.02 ml/cm2.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: CGF injection — CGF injection subdermally to expanded skin at the density of 0.02ml/cm2.
  Arms: CGF injection group
Procedure: Control — Saline will be injected into expanded skin
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluating whether autologous Concentrate Growth Factors(CGF) is safe and/or effective to accelerating skin regeneration and soft tissue expansion.

ELIGIBILITY:
Inclusion Criteria:

* Age of 14 to 65 years;
* Expanding skin donor site at the face, neck, anterior chest wall, abdominal wall or back;
* Persistent high level of expander internal pressure;
* Need for further skin expansion;

Exclusion Criteria:

* • Not fit for soft tissue expansion treatment;

  * Evidence of infection, ischemia, ulcer or other pathological changes within the targeting area which defined as not suitable for expansion; or history of delayed healing, radiational therapy;
  * Significant renal, cardiovascular, hepatic and psychiatric diseases;
  * Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV)
  * BMI >30;
  * History of any hematological disease, including leukopenia , thrombocytopenia, or thrombocytosis;
  * History of allogenic bone marrow transplantation;
  * Long history of smoking;
  * Evidence of malignant diseases or unwillingness to participate.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
To Measure the Change in Inflation Volume of the Silicone Expander From Baseline at 8 Weeks | baseline and 8 weeks post treatment
  Record the inflation volume(ml) of each expander with the maintained inner pressure. The inflation volume was recorded according to the injection volume during expansion.

SECONDARY OUTCOMES:
To Measure the Texture of Expanded Flap With Canfield's Visia Scanner | baseline and 8 weeks post treatment
  Evaluate skin texture with Canfield's Visia skin analysis imaging system and compare the characteristics including RBX red, RBX brown, pores, spots, et al.
Occurence of Major Adverse Events | Up to approximately 24 months after study start
  Including expanded flap ischaemia, necrosis, fluidify, infection, and all other adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided